CLINICAL TRIAL: NCT07227272
Title: Enhancing the Accuracy of Self-Reported Dietary Intake in Young Children: Development of Two Proxy Reporting Protocols for Self-Reported Dietary Assessment
Brief Title: Early Childhood Dietary Assessment Study
Acronym: ECDAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Executive Associate Dean of Research & Operations, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UTK IRB-25-08725-XP
Record Dates: First submitted 2025-06-30; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dietary Assessment
Keywords: Dietary Assessment; Assessment; Nutrition; Children
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional 24HR (Active Comparator): Caregivers will be asked to provide study-provided foods to their child and complete a traditional 24-hour dietary recall using the USDA five-step multiple-pass method.
  Interventions: Other: Traditional 24-hour dietary recall
- EMA-Assisted 24HR (Experimental): In the EMA+24HR condition, caregivers will receive study-provided foods for one meal and two snacks for three consecutive days. Caregivers will receive information on accessing an online EMA platform, and will be asked to upload pre- and post-photographs of the foods that their child eats over the three days. Additionally, any caregiver with whom the child consumes food outside of the primary proxy reporter will be trained by the primary caregiver and will be given access to upload photographs to the EMA site. The day following consumption of study-provided food, the caregiver will complete a 24HR using the USDA 5-step multiple-pass method by a trained research assistant. The research assistant will have access to all pre- and post-photographs and will prompt the caregiver for misreporting related to the photographs uploaded (i.e., time misreporting, omissions, intrusions, description, and amount misreporting).
  Interventions: Other: Ecological Momentary Assessment

INTERVENTIONS:
Other: Ecological Momentary Assessment — The EMA platform will allow for the primary caregiver (or any other adult with whom the child eats foods with) to upload pre- and post-photographs of all eating occasions. The photographs will be time-stamped and will be used by trained research assistants during the 24HR to aid in collection of accurate information about what the child consumed. The research assistant will be trained on how to prompt the caregiver for inaccuracies in reporting as needed.
  Arms: EMA-Assisted 24HR
Other: Traditional 24-hour dietary recall — Participants will complete a traditional 24-hour dietary recall via telephone, following the USDA five-step multiple pass method. Participants will receive a standardized food amounts booklet (FAB) to help with quantifying portion sizes consumed.
  Arms: Traditional 24HR

SUMMARY:
The goal of this crossover randomized controlled trial is to develop a proxy reporting protocol for a traditional 24-hour dietary recall (24HR) and an ecological momentary assessment (EMA) assisted 24-HR for use among children between the ages of 2 and 5 years. The main aims are to:

1. Assess the usability and feasibility of each proxy-reporting protocol and dietary assessment methodology.
2. Describe the dietary misreporting captured using each proxy-reporting protocol, and
3. Explore the accuracy of energy intake estimation of the 24HR and EMA+24HR methods, compared to objectively measured food intake.

During the research study, participants will:

1. Be provided with one meal and two snacks each day to provide to their child on three consecutive days. Foods can be offered to their child at times of their choosing, and leftovers will be placed back into reusable food storage containers to be picked up by research study staff. Uneaten foods will be weighed for an objective measure of intake.
2. The day after study-provided foods are given to the child, the adult caregiver will complete a proxy-reported 24HR phone call with a trained research assistant.
3. In the EMA+24HR condition, caregivers will be provided access to an online platform where they will upload pre- and post-photographs of all of their child's eating occasions across the three days that study-provided foods are eaten.

DETAILED DESCRIPTION:
This crossover, randomized controlled trial compares two proxy-reported dietary assessment protocols among caregivers with a child between the ages of 2 and 5 years. It also examines the dietary misreporting captured in each protocol and the accuracy of energy intake estimation from each methodology compared to objectively measured food intake. Caregivers with a child between the ages of 2 and 5 years and randomly assigned to one of two starting conditions: 1) traditional 24-hour dietary recall (24HR) or 2) Ecological momentary assessment (EMA)-assisted 24HR (EMA+24HR). Caregivers will complete the first assessment condition, and then, following a two-week washout period, will complete the other condition. In both conditions, caregivers will receive one meal and two snacks to provide to their child on three consecutive days. In addition to providing food, caregivers will identify a second caregiver (i.e., another parent, adult sibling, outside family member, or childcare worker) who will provide at least two eating occasions with study-provided foods over the three days. Including a caregiver outside of the primary proxy reporter will help assess the ability to accurately capture foods consumed away from the primary reporter, which has been identified as a challenge in dietary assessment among young children. The day after the child consumes study-provided foods, the caregiver will complete a 24HR via telephone with a trained research assistant following the United States Department of Agriculture five-step multiple pass method. After completing each dietary assessment condition, caregivers will complete an electronic survey that assesses the usability and acceptability of each proxy reporting protocol and dietary assessment condition.

The primary aims of this study are to:

1. Assess the feasibility, which will include the usability and acceptability, of the proxy reporting protocol for the 24HR and EMA+24HR.
2. Describe the dietary misreporting captured in the 24HR and EMA+24HR assessment strategies.

A secondary aim of the study will be to explore the accuracy, via determining agreement, of the 24 and EMA+24HR methods compared to objectively measured food intake, specifically in regard to energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregiver ≥ 18 years old
* Absence of food allergies or dietary restrictions for medical reasons (for the child)
* Caregiver reports child likes at least 70% of the study-provided foods from the pre-defined list of food options
* Caregiver has access to a smartphone device compatible with the EMA platform
* Caregiver can identify a second adult caregiver with access to a smartphone device compatible with the EMA platform and willing to provide the child with study-provided foods for at least two eating occasions.

Exclusion Criteria:

* Caregiver unwilling to feed study-provided foods to their child
* Caregiver unwilling to take pre-and-post photos of child's eating occasions
* Caregiver unwilling or unable to identify a second adult caregiver meeting the eligibility criteria
* Caregiver and child reside in a separate household for > 2 days per week
* Family resides >25 miles outside of the Knoxville, Tennessee, metropolitan area.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Usability - EMA+24HR Proxy-Reporting Protocol | Upon completion of the EMA+24HR condition
  Usability of the proxy-reporting protocol for the EMA+24HR condition will be assessed using a self-reported questionnaire. Survey items will focus on adequacy of training and support received, experience communicating with other caregivers regarding what children consumed when they weren't with them, and experience completing the proxy-reported 24HR.
Acceptability - EMA+24HR Proxy-Reporting Protocol | Upon completion of the EMA+24HR condition
  Acceptability of the proxy-reporting protocol for the EMA+24HR condition will be assessed using a self-reported questionnaire. Survey items will focus on caregivers' satisfaction with training and support received, their experience communicating with other caregivers regarding what children consumed when they weren't with them, their experience completing the proxy-reported 24HR, and overall satisfaction.
Usability of EMA Online Platform | Upon completion of the EMA+24HR condition
  Usability of the online EMA platform will be assessed by comparing the number of pre- and post-photos collected to the self-reported eating occasions captured in the proxy-reported 24HR.
Usability - Interface of EMA Platform | Upon completion of the EMA+24HR condition
  The usability of the online EMA interface will be assessed using a self-report questionnaire by using the usefulness and interface quality subscales from the Post-Study System Usability Questionnaire.
Acceptability - Online EMA Platform | Upon completion of the EMA+24HR condition
  Four items from the Theoretical Framework of Acceptability (TFA) measure will be used to assess acceptability of the EMA platform, focusing on four constructs 1) affective attitudes, 2) burden, 3) self-efficacy, and 4) general acceptability.
Usability - Traditional 24HR Proxy-Reporting Protocol | Upon completion of the traditional 24HR condition
  Usability of proxy-reporting protocols for the traditional 24HR condition will be assessed using a self-reported questionnaire. Survey items will focus on adequacy of training and support received, experience communicating with other caregivers regarding what children consumed when they weren't with them, and experience completing the proxy-reported 24HR.
Acceptability - Traditional 24HR Proxy Reporting Protocol | Upon completion of the traditional 24HR condition
  Acceptability of the proxy-reporting protocol for the traditional 24HR condition will be assessed using a self-reported questionnaire. Survey items will focus on caregivers' satisfaction with training and support received, their experience communicating with other caregivers regarding what children consumed when they weren't with them, their experience completing the proxy-reported 24HR, and overall satisfaction.
Dietary Misreporting - EMA+24HR Condition | Upon completion of the EMA+24HR condition
  Frequency of dietary misreporting (i.e., time-misreporting, omissions, intrusions, description and amount misreporting) will be assessed in the EMA+24HR by comparison of self-reported dietary assessment to photos uploaded to the EMA platform.
Dietary Misreporting - Traditional 24HR Condition | Upon completion of the traditional 24HR condition.
  Frequency of omissions will be assessed in the traditional 24HR condition using pre-post food weights to proxy-reported intake from the primary caregiver.

SECONDARY OUTCOMES:
Accuracy of Energy Intake Estimation - EMA+24HR Condition | Upon completion of EMA+24HR Condition
  The accuracy of the EMA+24HR condition will be assessed by comparing self-reported estimation of study-provided foods obtained from proxy-reporters with objectively measured food intake (pre-post food weights).
Accuracy of Energy Intake Estimation - Traditional Condition | Upon completion of the Traditional 24HR condition
  The accuracy of the traditional condition will be assessed by comparing self-reported estimation of study-provided foods obtained from proxy-reporters with objectively measured food intake (pre-post food weights).

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Lab, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Reilly JJ, Montgomery C, Jackson D, MacRitchie J, Armstrong J. Energy intake by multiple pass 24 h recall and total energy expenditure: a comparison in a representative sample of 3-4-year-olds. Br J Nutr. 2001 Nov;86(5):601-5. doi: 10.1079/bjn2001449. PMID 11737958
- [Background] Wallace A, Kirkpatrick SI, Darlington G, Haines J. Accuracy of Parental Reporting of Preschoolers' Dietary Intake Using an Online Self-Administered 24-h Recall. Nutrients. 2018 Jul 29;10(8):987. doi: 10.3390/nu10080987. PMID 30060605
- [Background] Bornhorst C, Huybrechts I, Ahrens W, Eiben G, Michels N, Pala V, Molnar D, Russo P, Barba G, Bel-Serrat S, Moreno LA, Papoutsou S, Veidebaum T, Loit HM, Lissner L, Pigeot I; IDEFICS consortium. Prevalence and determinants of misreporting among European children in proxy-reported 24 h dietary recalls. Br J Nutr. 2013 Apr 14;109(7):1257-65. doi: 10.1017/S0007114512003194. Epub 2012 Aug 6. PMID 22863030
- [Background] Livingstone MB, Robson PJ. Measurement of dietary intake in children. Proc Nutr Soc. 2000 May;59(2):279-93. doi: 10.1017/s0029665100000318. PMID 10946797
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Food and Nutrition Board; Callahan EA, editor. Approaches to Assessing Intake of Food and Dietary Supplements in Pregnant Women and Children 2 to 11 Years of Age: Proceedings of a Workshop Series. Washington (DC): National Academies Press (US); 2022 Jan 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK576562/ PMID 35041355
- [Background] Ravelli MN, Schoeller DA. Traditional Self-Reported Dietary Instruments Are Prone to Inaccuracies and New Approaches Are Needed. Front Nutr. 2020 Jul 3;7:90. doi: 10.3389/fnut.2020.00090. eCollection 2020. PMID 32719809